CLINICAL TRIAL: NCT03721978
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of VGX-3100 Delivered Intramuscularly Followed by Electroporation With CELLECTRA™ 5PSP for the Treatment of HPV-16 and/or HPV-18 Related High Grade Squamous Intraepithelial Lesion (HSIL) of the Cervix
Brief Title: REVEAL 2 Trial (Evaluation of VGX-3100 and Electroporation for the Treatment of Cervical HSIL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPV-303; 2018-004114-17 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cervical Dysplasia; Cervical High Grade Squamous Intraepithelial Lesion; HSIL
Keywords: Cervical intraepithelial neoplasia (CIN); CIN 2; CIN 3; Human papillomavirus (HPV); HPV-16; HPV-18; High Grade Squamous Intraepithelial Lesion (HSIL); papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions | interventions — VGX-3100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VGX-3100 + EP (Experimental): Participants received 3 IM injections of 6 mg (in 1 mL) VGX-3100 followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
  Interventions: Biological: VGX-3100; Device: CELLECTRA™-5PSP
- Matched Placebo + EP (Placebo Comparator): Participants received 3 IM injections of 1 mL VGX-3100 matching placebo followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
  Interventions: Biological: Matched Placebo; Device: CELLECTRA™-5PSP

INTERVENTIONS:
Biological: VGX-3100 — 1 milliliter (mL) VGX-3100 injected IM.
  Arms: VGX-3100 + EP
Biological: Matched Placebo — 1 mL of matched Placebo injected IM.
  Arms: Matched Placebo + EP
Device: CELLECTRA™-5PSP — CELLECTRA™-5PSP used for EP following IM injection of VGX 3100.

SUMMARY:
HPV-303 is a prospective, randomized, double-blind, placebo-controlled study of VGX-3100 delivered intramuscularly (IM) followed by electroporation (EP) delivered with CELLECTRA™ 5PSP in adult women with histologically confirmed high-grade squamous intraepithelial lesions (HSIL) (cervical intraepithelial neoplasia grade 2 [CIN2] or grade 3 [CIN3]) of the cervix, associated with human papillomavirus (HPV-16) and/or HPV-18.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and above
* Confirmed cervical infection with HPV types 16 and/or 18 at screening
* Cervical tissue specimen/slides provided to Study Pathology Adjudication Committee for diagnosis scheduled to be collected within 10 weeks prior to anticipated date of first dose of study drug
* Confirmed histologic evidence of cervical HSIL at screening
* Must be judged by Investigator to be an appropriate candidate for the protocol-specified procedure required at Week 36
* With respect to their reproductive capacity must be post-menopausal or surgically sterile or willing to use a contraceptive method with failure rate of less than 1% per year when used consistently and correctly from screening until Week 36
* Normal screening electrocardiogram (ECG)

Exclusion Criteria:

* Microscopic or gross evidence of adenocarcinoma-in-situ (AIS), high grade vulvar, vaginal, or anal intraepithelial neoplasia or invasive cancer in any histopathologic specimen at screening
* Cervical lesion(s) that cannot be fully visualized on colposcopy
* History of endocervical curettage (ECC) which showed cervical HSIL indeterminate, or insufficient for diagnosis
* Treatment for cervical HSIL within 4 weeks prior to screening
* Pregnant, breastfeeding or considering becoming pregnant during the study
* History of previous therapeutic HPV vaccination
* Immunosuppression as a result of underlying illness or treatment
* Receipt of any non-study, non-live vaccine within 2 weeks of Day 0
* Receipt of any non-study, live vaccine within 4 weeks of Day 0
* Current or history of clinically significant, medically unstable disease or condition which, in the judgment of the investigator, would jeopardize the safety of the participant, interfere with study assessments or endpoint evaluation, or otherwise impact the validity of the study results
* Presence of acute or chronic bleeding or clotting disorder that would contraindicate IM injections, or use of blood thinners within 2 weeks of Day 0
* Participation in an interventional study with an investigational compound or device within 30 days of signing informed consent
* Less than two acceptable sites available for IM injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 203 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (53):
- United States (27):
  - Visions Clinical Research- Tucson, Tucson, Arizona
  - Nuvance Health, Danbury, Connecticut
  - Christiana Care Health System, Newark, Delaware
  - Altus Research, Lake Worth, Florida
  - Salom and Tangir LLC, Miramar, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Augusta University, Augusta, Georgia
  - Affinity Clinical Research Institute, Oak Brook, Illinois
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Unified Women's Clinical Research - Hagerstown, Hagerstown, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Saginaw Valley Medical Research Group LLC, Saginaw, Michigan
  - Meridian Clinical Research Norfolk, Norfolk, Nebraska
  - New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Suffolk Obstetrics and Gynecology, Port Jefferson, New York
  - Montefiore Medical Center, The Bronx, New York
  - Unified Women's Clinical Research - Greensboro, Greensboro, North Carolina
  - Unified Women's Clinical Research - Morehead City, Morehead City, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - ClinOhio Research Services, Columbus, Ohio
  - Obstetrics & Gynecology Associates, Inc., Fairfield, Ohio
  - Frontier Clinical Research-Smithfield, Smithfield, Pennsylvania
  - Venus Gynecology, LLC, Myrtle Beach, South Carolina
  - Women's Physician Group Suite 203, Memphis, Tennessee
  - Storks Research, Sugar Land, Texas
  - Group For Women - Tidewater Clinical Research Inc., Virginia Beach, Virginia
- Argentina (3):
  - Instituto de Ginecología, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - DIM Clinica Privada, Ramos Mejía
- Brazil (5):
  - Associação Obras Sociais Irmã Dulce Hospital Santo Antônio, Salvador, Estado de Bahia
  - Hospital das Clinicas de Goiânia, Goiânia, Goiás
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
- Estonia (3):
  - Pärnu Hospital, Pärnu, Pärnumaa
  - East Tallinn Central Hospital Womens Clinic, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - HUS Naistentaudit ja synnytykset, Helsinki, Uusimaa
  - Northern Savo Hospital District Muncipal Federation, Kuopio
- Lithuania (2):
  - Vilnius District Central Outpatient Clinic, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (3):
  - Niepubliczny Zakład Opieki Zdrowotnej Profimed, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin, Lublin Voivodeship
  - Centrum Medyczne Angelius Provita, Śląskie
- Puerto Rico Translational Research Center (PRTRC), Rio Piedras, Puerto Rico
- South Africa (2):
  - Lynette Reynders Private Practice, Centurion, Gauteng
  - University of Cape Town, Cape Town, Western Cape
- Spain (5):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 53 study sites from 28 February 2019 to 15 September 2022.
Pre-assignment Details: A total of 203 participants with human papillomavirus (HPV)-16 and/or HPV-18 related high-grade squamous intraepithelial lesion (HSIL) of the cervix were randomized in 2:1 to receive either VGX-3100+Electroporation (EP) or Matched Placebo+EP.
Groups:
- VGX-3100 + EP: Participants received 3 intramuscular (IM) injections of 6 milligram (mg) (in 1 milliliter [mL]) VGX-3100 followed by EP using the CELLECTRA™-5PSP device on Day 0, Week 4, and Week 12.
Period: Overall Study
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Started | 134 | 69
Intent-to-Treat (ITT) Population (ITT population included all participants who were randomized.) | 134 | 69
Baseline Biomarker-positive Participants for ITT (Baseline Biomarker-positive Participants for ITT included participants from ITT population who were biomarker positive as identified by microRNA (miRNA) profiling performed from peripheral blood.) | 21 | 4
Safety Set (Safety set included all participants who received at least one dose of study treatment.) | 134 | 68
Modified ITT (mITT) Population (mITT population included all participants who received at least one dose of study treatment and who had an analysis endpoint of interest.) | 130 | 68
Completed | 121 | 64
Not Completed | 13 | 5
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Progressive Disease | 1 | 0
Not completed — Lost to Follow-up | 5 | 1
Not completed — Reason not Specified | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | VGX-3100 + EP | Matched Placebo + EP | Total
Number analyzed (Participants) | 134 | 69 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (6.98) | 31.1 (7.93) | 31.4 (7.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 69 | 203
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 16 | 41
  Not Hispanic or Latino | 108 | 53 | 161
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 3
  Black or African American | 8 | 2 | 10
  White | 116 | 66 | 182
  Other | 2 | 0 | 2
  Multiple | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Histologic Evidence of Cervical HSIL on Histology Sample and No Evidence of HPV-16 and/or HPV-18 in Cervical Samples
Description: Baseline biomarker-positive participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL, no evidence of HPV-16 and/or HPV-18 at Week 36, and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or low-grade intraepithelial lesion (LSIL). Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep™. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized. Only baseline biomarker-positive participants were planned to be analyzed for this outcome measure. Baseline Biomarker-positive Participants for ITT included participants from ITT population who were biomarker-positive as identified by miRNA profiling performed from peripheral blood.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 28.6 | 0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Superiority — Superiority was concluded if the one-sided p-value was <0.025 and the corresponding lower bound of the 95% CI exceeded zero (0); p = 0.115, Miettinen and Nurminen method; Difference in Percentage = 28.6, 95% CI 2-sided [-24.6 to 50.4]

2. Secondary Outcome: Baseline Biomarker-positive Participants for Safety Population: Number of Participants With Any Local and Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as AEs. Nausea, fatigue, injection site bruising, injection site erythema, injection site haematoma, injection site induration, injection site pain, injection site pruritus, injection site swelling, malaise, pyrexia, arthralgia, myalgia, headache and erythema were considered as local and systemic AEs for baseline biomarker-positive participants for safety population.
Time Frame: From Baseline to Week 40
Population: Safety set included all participants who received at least one dose of study treatment. Only baseline biomarker-positive participants were planned to be analyzed for this outcome measure. Baseline Biomarker-positive Participants for the safety set included participants from the safety set who were biomarker-positive as identified by miRNA profiling performed from peripheral blood.
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
Participants
  Nausea | 6 | 0
  Fatigue | 10 | 2
  Injection Site Bruising | 7 | 1
  Injection Site Erythema | 4 | 2
  Injection Site Haematoma | 1 | 0
  Injection Site Induration | 1 | 0
  Injection Site Pain | 19 | 4
  Injection Site Pruritus | 7 | 2
  Injection Site Swelling | 10 | 2
  Malaise | 2 | 1
  Pyrexia | 4 | 0
  Arthralgia | 6 | 0
  Myalgia | 13 | 2
  Headache | 13 | 3
  Erythema | 1 | 0

3. Secondary Outcome: Safety Population: Number of Participants With Local and Systemic AEs
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as AEs. Nausea, chills, fatigue, injection site bruising, injection site erythema, injection site haematoma, injection site haemorrhage, injection site induration, injection site oedema, injection site pain, injection site paraesthesia, injection site pruritus, injection site swelling, malaise, pain, pyrexia, temperature regulation disorder, arthralgia, myalgia, headache and erythema were considered as local and systemic AEs for safety population.
Time Frame: From Baseline to Week 40
Population: Safety set included all participants who received at least one dose of study treatment. 1 participant received mixed treatment in error. Safety data for this participant has been presented in a separate arm.
Measure: Count of Participants; unit: Participants
Groups:
- Mixed Treatment: Participant received one IM injection of 6 mg (in 1 mL) VGX-3100 on Day 0 followed by EP using the CELLECTRA™-5PSP device and 2 IM injections of 1 mL VGX-3100 matching placebo followed by EP using the CELLECTRA™-5PSP device on Week 4, and Week 12.
Arm/Group | VGX-3100 + EP | Matched Placebo + EP | Mixed Treatment
Number analyzed (Participants) | 134 | 67 | 1
Participants
  Nausea | 36 | 17 | 0
  Chills | 2 | 1 | 0
  Fatigue | 56 | 33 | 1
  Injection Site Bruising | 21 | 11 | 0
  Injection Site Erythema | 36 | 15 | 0
  Injection Site Haematoma | 10 | 7 | 0
  Injection Site Haemorrhage | 1 | 0 | 0
  Injection Site Induration | 3 | 0 | 0
  Injection Site Oedema | 5 | 2 | 0
  Injection Site Pain | 123 | 58 | 1
  Injection Site Paraesthesia | 1 | 0 | 0
  Injection Site Pruritus | 33 | 22 | 0
  Injection Site Swelling | 43 | 19 | 0
  Malaise | 18 | 12 | 1
  Pain | 1 | 1 | 0
  Pyrexia | 11 | 5 | 0
  Temperature Regulation Disorder | 1 | 0 | 0
  Arthralgia | 29 | 14 | 0
  Myalgia | 56 | 29 | 0
  Headache | 66 | 37 | 0
  Erythema | 1 | 0 | 0

4. Secondary Outcome: Baseline Biomarker-positive Participants for Safety Population: Number of Participants With Any Treatment Emergent AEs (TEAEs) and Serious TEAEs (Including Suspected Unexpected Serious Adverse Reaction [SUSAR] and Unexpected Adverse Device Effect [UADE])
Description: AE is any untoward medical occurrence in a participant administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. Serious AE (SAE) is any experience that suggested significant hazard, contraindication, side effect/precaution, & fulfilled any of the following: fatal, life-threatening, required in-patient hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant/required intervention to prevent other outcomes. TEAEs are any AEs starting on or after the first administration of any investigational product (IP). TEAEs included both serious and non-serious TEAEs. UADE is any SAE on health/safety or any life-threatening problem/death caused by, or associated with a device, if that effect, problem/death was not previously identified in nature, severity/degree of incidence in the investigational plan or application.
Time Frame: From Baseline to Week 40
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
Participants
  Participants with any TEAEs | 20 | 4
  Participants with any Serious TEAEs | 3 | 0
  Participants with SUSAR | 0 | 0
  Participants with UADE | 0 | 0

5. Secondary Outcome: Safety Population: Number of Participants With Any TEAEs and Serious TEAEs (Including SUSAR and UADE)
Description: AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. SAE is any experience that suggested significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal, life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent other outcomes. TEAEs are defined as AEs starting on or after the first administration of any IP. TEAEs included both serious and non-serious TEAEs. UADE is any SAE on health/safety or any life-threatening problem/death caused by, or associated with a device, if that effect, problem/death was not previously identified in nature, severity/degree of incidence in the investigational plan or application.
Time Frame: From Baseline to Week 40
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP | Mixed Treatment
Number analyzed (Participants) | 134 | 67 | 1
Participants
  Participants with any TEAEs | 131 | 67 | 1
  Participants with any Serious TEAEs | 9 | 9 | 0
  Participants with SUSAR | 0 | 0 | 0
  Participants with UADE | 0 | 0 | 0

6. Secondary Outcome: ITT Population: Percentage of Participants With No Histologic Evidence of Cervical HSIL on Histology Sample and No Evidence of HPV-16 and/or HPV-18 in Cervical Samples
Description: Participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL, no evidence of HPV-16 and/or HPV-18 at Week 36, and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or low-grade intraepithelial lesion (LSIL). Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep™. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 27.6 | 8.7
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, Miettinen and Nurminen method; Difference in Percentage = 18.9, 95% CI 2-sided [7.8 to 28.6]

7. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Histologic Evidence of Cervical HSIL on Histology Sample
Description: Baseline biomarker-positive participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL at Week 36 and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized. Only baseline biomarker-positive participants were planned to be analyzed for this outcome measure. Baseline Biomarker-positive Participants for ITT included participants from the ITT population who were biomarker-positive as identified by miRNA profiling performed from peripheral blood.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 38.1 | 25.0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 13.1, 95% CI 2-sided [-37.7 to 46.0]

8. Secondary Outcome: ITT Population: Percentage of Participants With No Histologic Evidence of Cervical HSIL on Histology Sample
Description: Participants with no histologic (i.e., biopsies or excisional treatment) evidence of cervical HSIL at Week 36 and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 34.3 | 21.7
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 12.6, 95% CI 2-sided [-0.8 to 24.5]

9. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Evidence of HPV-16 and/or HPV-18 in Cervical Samples by Type Specific HPV Testing
Description: Baseline biomarker-positive participants with no evidence of HPV-16 and/or HPV-18 at Week 36 time frame and participants in whom an excision or biopsy sample was not obtained between the initial dose up to Week 36 were considered to be responders. Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep™. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 38.1 | 0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 38.1, 95% CI 2-sided [-15.7 to 59.5]

10. Secondary Outcome: ITT Population: Percentage of Participants With No Evidence of HPV-16 and/or HPV-18 in Cervical Samples by Type Specific HPV Testing
Description: Participants with no evidence of HPV-16 and/or HPV-18 at Week 36 and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. Cervical samples for HPV-16 and/or HPV-18 were collected using the ThinPrep™. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 38.1 | 10.1
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 27.9, 95% CI 2-sided [16.0 to 38.2]

11. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Histologic Evidence of LSIL or HSIL on Histology Sample
Description: Baseline biomarker-positive participants with no histologic evidence of cervical HSIL, squamous atypia, or LSIL at Week 36 and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of LSIL was defined as no evidence of cervical squamous intraepithelial neoplasia 1 (CIN1), CIN2, or CIN3 on biopsies or excisional treatment. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 38.1 | 25.0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 13.1, 95% CI 2-sided [-37.7 to 46.0]

12. Secondary Outcome: ITT Population: Percentage of Participants With No Evidence of Histologic LSIL or HSIL on Histology Sample
Description: Participants with no histologic evidence of cervical HSIL, squamous atypia, or LSIL at Week 36 and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of LSIL was defined as no evidence of CIN1, CIN2, or CIN3 on biopsies or excisional treatment. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 32.1 | 14.5
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 17.6, 95% CI 2-sided [5.2 to 28.5]

13. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Evidence of LSIL or HSIL on Histology Sample and No Evidence of HPV-16 and/or HPV-18 by Type Specific HPV Testing
Description: Baseline biomarker-positive participants with no histologic evidence of cervical HSIL, squamous atypia, or LSIL, no evidence of HPV-16 and/or HPV-18 by type specific HPV testing at Week 36, and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of LSIL was defined as no evidence of CIN1, CIN2, or CIN3 on biopsies or excisional treatment. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 28.6 | 0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 28.6, 95% CI 2-sided [-24.6 to 50.4]

14. Secondary Outcome: ITT Population: Percentage of Participants With No Evidence of LSIL or HSIL on Histology Sample and No Evidence of HPV-16 and/or HPV-18 by Type Specific HPV Testing
Description: Participants with no histologic evidence of cervical HSIL, squamous atypia, or LSIL, no evidence of HPV-16 and/or HPV-18 by type specific HPV testing at Week 36, and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. No evidence of LSIL was defined as no evidence of CIN1, CIN2, or CIN3 on biopsies or excisional treatment. No evidence of HSIL was defined by histology as negative, squamous atypia, or LSIL. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: At Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 26.1 | 5.8
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 20.3, 95% CI 2-sided [10.1 to 29.5]

15. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants With No Progression of Cervical HSIL to Cervical Carcinoma
Description: Baseline biomarker-positive participants with no histologic evidence of cervical adenocarcinoma in situ (AIS) or cervical carcinoma at Week 36 relative to baseline and participants in whom an excision or biopsy sample was not obtained between initial dose up to Week 36 were considered as responders. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: From Baseline at Week 36
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 76.2 | 75.0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 1.2, 95% CI 2-sided [-31.2 to 50.5]

16. Secondary Outcome: ITT Population: Percentage of Participants With No Progression of Cervical HSIL to Cervical Carcinoma
Description: Participants with no histologic evidence of cervical AIS or cervical carcinoma at Week 36 relative to baseline and participants who did not have unscheduled excision or biopsy sample obtained between the initial dose up to Week 36 were considered to be responders. The efficacy time frame is defined by a biopsy or surgical excision at any time starting from 14 days prior to the protocol-specified target date of Week 36. The first tissue removal sample within the time frame determines the histology endpoint.
Time Frame: From Baseline at Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 82.1 | 76.8
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 5.3, 95% CI 2-sided [-6.0 to 17.9]

17. Secondary Outcome: Baseline Biomarker-positive Participants for ITT Population: Percentage of Participants Who Have Cleared HPV-16 and/or HPV-18 in Non-cervical Anatomic Locations
Description: Percentage of baseline biomarker-positive participants who have cleared HPV-16 and/or HPV-18 on specimens from non-cervical anatomic locations (oropharynx, vagina and intra-anal) at Week 36 Visit compared to baseline were reported.
Time Frame: From Baseline at Week 36
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 21 | 4
percentage of participants | 19.0 | 25.0
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = -6.0, 95% CI 2-sided [-54.7 to 25.8]

18. Secondary Outcome: ITT Population: Percentage of Participants Who Have Cleared HPV-16 and/or HPV-18 in Non-cervical Anatomic Locations
Description: Percentage of participants who have cleared HPV-16 and/or HPV-18 on specimens from non-cervical anatomic locations (oropharynx, vagina, and intra-anal) at Week 36 Visit compared to baseline were reported.
Time Frame: From Baseline at Week 36
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 134 | 69
percentage of participants | 22.4 | 10.1
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Test type: Other; Difference in Percentage = 12.2, 95% CI 2-sided [1.1 to 21.9]

19. Secondary Outcome: Baseline Biomarker-positive Participants for mITT Population: Serum Concentrations of Anti-HPV-16 and Anti-HPV-18 Antibody
Description: A standardized binding enzyme-linked immunosorbent assay (ELISA) was performed to measure the anti-HPV-16/18 antibody response induced by VGX-3100. E7 is a viral protein produced by cells infected by HPV-16/18.
Time Frame: At Week 15 and Week 36
Population: mITT population included all participants who received at least one dose of study treatment and who had analysis endpoint of interest. Baseline Biomarker-positive Participants for mITT included participants from the mITT population who were biomarker-positive as identified by miRNA profiling performed from peripheral blood. Overall number of participants analyzed is the number of participants with data available for this outcome measure.
Measure: Median (Full Range); unit: reciprocal endpoint titer
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 20 | 3
reciprocal endpoint titer
  HPV-16 E7 at Week 15 | 450.0 [1 to 18225] | 1.0 [1 to 1]
  HPV-16 E7 at Week 36 | 13.0 [1 to 18225] | 1.0 [1 to 18225]
  HPV-18 E7 at Week 15 | 4050.0 [1 to 18225] | 1.0 [1 to 1]
  HPV-18 E7 at Week 36 | 675.0 [1 to 18225] | 1.0 [1 to 18225]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 15: HPV-16 E7; Test type: Other; Location Shift = 449.0, 95% CI 2-sided [0.0 to 18224.0]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 36: HPV-16 E7; Test type: Other; Location Shift = 0.0, 95% CI 2-sided [-18224.0 to 674.0]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 15: HPV-18 E7; Test type: Other; Location Shift = 4049.0, 95% CI 2-sided [224.0 to 18224.0]
Statistical Analysis 4: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 36: HPV-18 E7; Test type: Other; Location Shift = 74.0, 95% CI 2-sided [-18000.0 to 6074.0]

20. Secondary Outcome: mITT Population: Serum Concentrations of Anti-HPV-16 and Anti-HPV-18 Antibody
Description: A standardized binding ELISA was performed to measure the anti-HPV-16/18 antibody response induced by VGX-3100. E7 is a viral protein produced by cells infected by HPV-16/18.
Time Frame: At Week 15 and Week 36
Population: mITT population included all participants who received at least one dose of study treatment and who had an analysis endpoint of interest. Overall number of participants analyzed is the number of participants with data available for this outcome measure. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Median (Full Range); unit: reciprocal endpoint titer
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 124 | 64
reciprocal endpoint titer
  HPV-16 E7 at Week 15 | 225.0 [1 to 18225] | 1.0 [1 to 75]
  HPV-16 E7 at Week 36: number analyzed (Participants) | 123 | 63
  HPV-16 E7 at Week 36 | 1.0 [1 to 18225] | 1.0 [1 to 18225]
  HPV-18 E7 at Week 15 | 2025.0 [1 to 18225] | 1.0 [1 to 18225]
  HPV-18 E7 at Week 36: number analyzed (Participants) | 123 | 63
  HPV-18 E7 at Week 36 | 675.0 [1 to 18225] | 1.0 [1 to 18225]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 15: HPV-16 E7; Test type: Other; Location Shift = 224.0, 95% CI 2-sided [224.0 to 674.0]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 36: HPV-16 E7; Test type: Other; Location Shift = 0.0, 95% CI 2-sided [0.0 to 24.0]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 15: HPV-18 E7; Test type: Other; Location Shift = 2024.0, 95% CI 2-sided [2024.0 to 6074.0]
Statistical Analysis 4: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Week 36: HPV-18 E7; Test type: Other; Location Shift = 674.0, 95% CI 2-sided [224.0 to 674.0]

21. Secondary Outcome: Baseline Biomarker-positive Participants for mITT Population: Change From Baseline in Interferon-Gamma Response Magnitude at Week 15 and 36
Description: Assessment of cellular immune activity occurred via the application of the Interferon-γ enzyme-linked immunosorbent spot (IFN-γ ELISpot). Peripheral blood mononuclear cells (PBMCs) isolated from whole blood sample were used for analysis. E6 and E7 are viral proteins produced by cells infected by HPV-16/18.
Time Frame: Baseline; Week 15 and Week 36
Population: mITT population=all participants who received at least one dose of study treatment and who had an analysis endpoint of interest. Baseline Biomarker-positive Participants for mITT=participants from mITT population who were biomarker-positive as identified by miRNA profiling performed from peripheral blood. Overall number analyzed=number of participants with data available for this outcome measure. Number analyzed=number of participants with data available for analysis at the specified timepoints.
Measure: Median (Full Range); unit: spot forming units (SFU)/10^6 PBMC
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 11 | 2
spot forming units (SFU)/10^6 PBMC
  HPV-16 E6: Baseline | 1.67 [0.0 to 11.7] | 4.17 [0.0 to 8.3]
  HPV-16 E6: Change from Baseline at Week 15: number analyzed (Participants) | 7 | 2
  HPV-16 E6: Change from Baseline at Week 15 | 25.00 [0.0 to 73.3] | 0.00 [0.0 to 0.0]
  HPV-16 E6: Change from Baseline at Week 36: number analyzed (Participants) | 6 | 1
  HPV-16 E6: Change from Baseline at Week 36 | 15.00 [0.0 to 38.3] | 0.0 [0.0 to 0.0]
  HPV-16 E7: Baseline | 0.00 [0.0 to 5.0] | 1.67 [0.0 to 3.3]
  HPV-16 E7: Change from Baseline at Week 15: number analyzed (Participants) | 7 | 2
  HPV-16 E7: Change from Baseline at Week 15 | 16.67 [0.0 to 85.0] | 0.00 [0.0 to 0.0]
  HPV-16 E7: Change from Baseline at Week 36: number analyzed (Participants) | 6 | 1
  HPV-16 E7: Change from Baseline at Week 36 | 5.00 [0.0 to 36.7] | 0.00 [0.0 to 0.0]
  HPV-18 E6: Baseline | 0.00 [0.0 to 11.7] | 2.50 [0.0 to 5.0]
  HPV-18 E6: Change from Baseline at Week 15: number analyzed (Participants) | 7 | 2
  HPV-18 E6: Change from Baseline at Week 15 | 26.67 [0.0 to 181.7] | 0.00 [0.0 to 0.0]
  HPV-18 E6: Change from Baseline at Week 36: number analyzed (Participants) | 6 | 1
  HPV-18 E6: Change from Baseline at Week 36 | 11.67 [0.0 to 31.7] | 0.00 [0.0 to 0.0]
  HPV-18 E7: Baseline | 0.00 [0.0 to 3.3] | 4.17 [0.0 to 8.3]
  HPV-18 E7: Change from Baseline at Week 15: number analyzed (Participants) | 7 | 2
  HPV-18 E7: Change from Baseline at Week 15 | 3.33 [0.0 to 46.7] | 0.00 [0.0 to 0.0]
  HPV-18 E7: Change from Baseline at Week 36: number analyzed (Participants) | 6 | 1
  HPV-18 E7: Change from Baseline at Week 36 | 4.17 [0.0 to 20.0] | 0.00 [0.0 to 0.0]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E6: Week 15; Test type: Other; Location Shift = 25.00, 95% CI 2-sided [0.00 to 73.33]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E6: Week 36; Test type: Other; Location Shift = 15.00, 95% CI 2-sided [0.00 to 38.33]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E7: Week 15; Test type: Other; Location Shift = 16.67, 95% CI 2-sided [0.00 to 85.00]
Statistical Analysis 4: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E7: Week 36; Test type: Other; Location Shift = 5.00, 95% CI 2-sided [0.00 to 36.67]
Statistical Analysis 5: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E6: Week 15; Test type: Other; Location Shift = 26.67, 95% CI 2-sided [0.00 to 181.67]
Statistical Analysis 6: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E6: Week 36; Test type: Other; Location Shift = 11.67, 95% CI 2-sided [0.00 to 31.67]
Statistical Analysis 7: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E7: Week 15; Test type: Other; Location Shift = 3.33, 95% CI 2-sided [0.00 to 46.67]
Statistical Analysis 8: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E7: Week 36; Test type: Other; Location Shift = 4.17, 95% CI 2-sided [0.00 to 20.00]

22. Secondary Outcome: mITT Population: Change From Baseline in Interferon-Gamma Response Magnitude at Week 15 and 36
Description: Assessment of cellular immune activity occurred via the application of the IFN-γ ELISpot. PBMCs isolated from whole blood sample were used for analysis. E6 and E7 are viral proteins produced by cells infected by HPV-16/18.
Time Frame: Baseline; Week 15 and Week 36
Population: mITT population included all participants who received at least one dose of clinical trial treatment and who had an analysis endpoint of interest. Overall number of participants analyzed is the number of participants with data available for this outcome measure. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Median (Full Range); unit: SFU/10^6 PBMC
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 92 | 51
SFU/10^6 PBMC
  HPV-16 E6: Baseline | 1.67 [0.0 to 25.0] | 0.00 [0.0 to 15.8]
  HPV-16 E6: Change from Baseline at Week 15: number analyzed (Participants) | 70 | 34
  HPV-16 E6: Change from Baseline at Week 15 | 10.00 [0.0 to 115.0] | 1.67 [0.0 to 16.7]
  HPV-16 E6: Change from Baseline at Week 36: number analyzed (Participants) | 66 | 41
  HPV-16 E6: Change from Baseline at Week 36 | 8.33 [0.0 to 110.0] | 0.00 [0.0 to 23.3]
  HPV-16 E7: Baseline | 0.00 [0.0 to 11.7] | 0.00 [0.0 to 15.0]
  HPV-16 E7: Change from Baseline at Week 15: number analyzed (Participants) | 70 | 34
  HPV-16 E7: Change from Baseline at Week 15 | 6.67 [0.0 to 236.7] | 0.00 [0.0 to 21.7]
  HPV-16 E7: Change from Baseline at Week 36: number analyzed (Participants) | 66 | 41
  HPV-16 E7: Change from Baseline at Week 36 | 3.33 [0.0 to 101.7] | 0.00 [0.0 to 8.3]
  HPV-18 E6: Baseline | 0.00 [0.0 to 11.7] | 0.00 [0.0 to 11.7]
  HPV-18 E6: Change from Baseline at Week 15: number analyzed (Participants) | 70 | 34
  HPV-18 E6: Change from Baseline at Week 15 | 26.67 [0.0 to 885.0] | 0.00 [0.0 to 68.3]
  HPV-18 E6: Change from Baseline at Week 36: number analyzed (Participants) | 66 | 41
  HPV-18 E6: Change from Baseline at Week 36 | 19.17 [0.0 to 510.0] | 0.00 [0.0 to 35.0]
  HPV-18 E7: Baseline | 0.00 [0.0 to 13.3] | 0.00 [0.0 to 18.3]
  HPV-18 E7: Change from Baseline at Week 15: number analyzed (Participants) | 70 | 34
  HPV-18 E7: Change from Baseline at Week 15 | 5.83 [0.0 to 291.7] | 0.00 [0.0 to 15.0]
  HPV-18 E7: Change from Baseline at Week 36: number analyzed (Participants) | 66 | 41
  HPV-18 E7: Change from Baseline at Week 36 | 3.33 [0.0 to 246.7] | 0.00 [0.0 to 135.0]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E6: Week 15; Test type: Other; Location Shift = 8.33, 95% CI 2-sided [3.33 to 11.67]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E6: Week 36; Test type: Other; Location Shift = 5.83, 95% CI 2-sided [3.33 to 11.67]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E7: Week 15; Test type: Other; Location Shift = 5.00, 95% CI 2-sided [1.67 to 11.67]
Statistical Analysis 4: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-16 E7: Week 36; Test type: Other; Location Shift = 1.67, 95% CI 2-sided [0.00 to 5.00]
Statistical Analysis 5: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E6: Week 15; Test type: Other; Location Shift = 25.00, 95% CI 2-sided [15.00 to 40.00]
Statistical Analysis 6: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E6: Week 36; Test type: Other; Location Shift = 16.67, 95% CI 2-sided [10.00 to 28.33]
Statistical Analysis 7: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E7: Week 15; Test type: Other; Location Shift = 3.33, 95% CI 2-sided [1.67 to 6.67]
Statistical Analysis 8: Comparison: VGX-3100 + EP vs Matched Placebo + EP; HPV-18 E7: Week 36; Test type: Other; Location Shift = 1.67, 95% CI 2-sided [0.00 to 3.33]

23. Secondary Outcome: Baseline Biomarker-positive Participants for mITT Population: Change From Baseline in Flow Cytometry Response Magnitude at Week 15
Description: Assessment of cellular immune activity was measured using the application flow cytometry for the purposes of performing a Lytic Granule Loading Assay. The Lytic Granule Loading assay examines the following external cellular markers: CD3, CD4, CD8 (T cell identification), CD137, CD38, and CD69 (T cell activation markers) as well as PD-1 (exhaustion/activation marker). Here, changes from baseline in the percentage of CD8+CD137+Perforin+, CD8+CD38+Perforin+, and CD8+CD69+Perforin+ are reported.
Time Frame: Baseline, Week 15
Population: Baseline Biomarker-positive Participants for mITT=participants from the mITT population who were biomarker-positive as identified by miRNA profiling performed from peripheral blood. Overall number of participants analyzed is the number of participants with data available for this outcome measure. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Median (Full Range); unit: percentage of cells
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 15 | 2
percentage of cells
  CD8+CD137+Perforin+: Baseline | 0.000 [0.00 to 0.16] | 0.020 [0.00 to 0.04]
  CD8+CD137+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 14 | 2
  CD8+CD137+Perforin+: Change from Baseline at Week 15 | 0.035 [0.00 to 0.33] | 0.002 [0.00 to 0.002]
  CD8+CD38+Perforin+: Baseline | 0.000 [0.00 to 0.04] | 0.027 [0.00 to 0.05]
  CD8+CD38+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 14 | 2
  CD8+CD38+Perforin+: Change from Baseline at Week 15 | 0.005 [0.00 to 0.21] | 0.000 [0.00 to 0.00]
  CD8+CD69+Perforin+: Baseline | 0.008 [0.00 to 0.05] | 0.003 [0.00 to 0.01]
  CD8+CD69+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 14 | 2
  CD8+CD69+Perforin+: Change from Baseline at Week 15 | 0.042 [0.00 to 0.31] | 0.030 [0.00 to 0.05]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD137+Perforin+; Test type: Other; Location Shift = 0.033, 95% CI 2-sided [-0.004 to 0.325]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD38+Perforin+; Test type: Other; Location Shift = 0.005, 95% CI 2-sided [0.000 to 0.208]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD69+Perforin+; Test type: Other; Location Shift = 0.014, 95% CI 2-sided [-0.055 to 0.310]

24. Secondary Outcome: mITT Population: Change From Baseline in Flow Cytometry Response Magnitude at Week 15
Description: as for outcome 23
Time Frame: Baseline, Week 15
Population: as for outcome 22
Measure: Median (Full Range); unit: percentage of cells
Arm/Group | VGX-3100 + EP | Matched Placebo + EP
Number analyzed (Participants) | 95 | 48
percentage of cells
  CD8+CD137+Perforin+: Baseline | 0.000 [0.00 to 0.29] | 0.012 [0.00 to 0.24]
  CD8+CD137+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 89 | 44
  CD8+CD137+Perforin+: Change from Baseline at Week 15 | 0.049 [0.00 to 0.33] | 0.000 [0.00 to 0.10]
  CD8+CD38+Perforin+: Baseline | 0.001 [0.00 to 0.09] | 0.007 [0.00 to 0.09]
  CD8+CD38+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 89 | 44
  CD8+CD38+Perforin+: Change from Baseline at Week 15 | 0.023 [0.00 to 0.27] | 0.000 [0.00 to 0.07]
  CD8+CD69+Perforin+: Baseline | 0.003 [0.00 to 0.14] | 0.007 [0.00 to 0.09]
  CD8+CD69+Perforin+: Change from Baseline at Week 15: number analyzed (Participants) | 89 | 44
  CD8+CD69+Perforin+: Change from Baseline at Week 15 | 0.037 [0.00 to 0.31] | 0.000 [0.00 to 0.06]
Statistical Analysis 1: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD137+Perforin+; Test type: Other; Location Shift = 0.041, 95% CI 2-sided [0.004 to 0.077]
Statistical Analysis 2: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD38+Perforin+; Test type: Other; Location Shift = 0.011, 95% CI 2-sided [0.003 to 0.028]
Statistical Analysis 3: Comparison: VGX-3100 + EP vs Matched Placebo + EP; Parameter: CD8+CD69+Perforin+; Test type: Other; Location Shift = 0.034, 95% CI 2-sided [0.022 to 0.053]

ADVERSE EVENTS:
Time Frame: From Baseline to Week 40
Description: Safety set included all participants who received at least one dose of study treatment. 1 participant received mixed treatment in error. Safety data for this participant has been presented in a separate arm.
Groups:
- Mixed Treatment: Participants received one IM injection of 6 mg (in 1 mL) VGX-3100 on Day 0 followed by EP using the CELLECTRA™-5PSP device and 2 IM injections of 1 mL VGX-3100 matching placebo followed by EP using the CELLECTRA™-5PSP device on Week 4, and Week 12.
Arm/Group | VGX-3100 + EP | Matched Placebo + EP | Mixed Treatment
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/67 | 0/1
Serious Adverse Events (participants affected / at risk) | 9/134 | 9/67 | 0/1
Other Adverse Events (participants affected / at risk) | 131/134 | 67/67 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + EP (N=134) | Matched Placebo + EP (N=67) | Mixed Treatment (N=1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Ovarian rupture (Reproductive system and breast disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 + EP (N=134) | Matched Placebo + EP (N=67) | Mixed Treatment (N=1)
Headache (Nervous system disorders) | 66 | 37 | 0
Dizziness (Nervous system disorders) | 8 | 2 | 0
Injection site pain (General disorders) | 123 | 58 | 1
Fatigue (General disorders) | 56 | 33 | 1
Injection site swelling (General disorders) | 43 | 19 | 0
Injection site erythema (General disorders) | 36 | 15 | 0
Injection site pruritus (General disorders) | 33 | 22 | 0
Injection site bruising (General disorders) | 21 | 11 | 0
Malaise (General disorders) | 18 | 12 | 1
Pyrexia (General disorders) | 11 | 5 | 0
Injection site haematoma (General disorders) | 10 | 7 | 0
Nausea (Gastrointestinal disorders) | 36 | 17 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 56 | 29 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 14 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
COVID-19 (Infections and infestations) | 12 | 8 | 0
Urinary tract infection (Infections and infestations) | 8 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03721978/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT03721978/SAP_001.pdf